CLINICAL TRIAL: NCT04737577
Title: Phase II Pilot Randomized Controlled Trial to Assess Feasibility of "Supra-marginal" Surgical Resection of Malignant Glioma
Brief Title: Glioma Supra Marginal Incision Trial
Acronym: G-SUMIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Sunnybrook Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CTO 3297
Record Dates: First submitted 2021-01-19; First posted 2021-02-04 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: High Grade Glioma
Keywords: Supramarginal resection; Standard total resection; Surgery; Brain tumor; HGG
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supramarginal resection (intervention arm) (Experimental): Planned resection beyond the Gadolinium (GAD)-enhancing region extending to either at least 1 cm into non-enhancing tissue, or the nearest non-enhancing sulcal boundary/ventricle wall if these structures are closer than 1 cm.
  Interventions: Procedure: Supramarginal resection
- Conventional (i.e. GTR) resection (Other): Planned resection of ≥95% of the GAD-enhancing regions of tumor without expanding the resection beyond this margin.
  Interventions: Procedure: Conventional (i.e. GTR) resection

INTERVENTIONS:
Procedure: Supramarginal resection — Tissue removal beyond the GAD-enhancing region extending to either at least 1 cm into non-enhancing tissue, or the nearest non-enhancing sulcal boundary/ventricle wall if these structures are closer than 1 cm.
  Arms: Supramarginal resection (intervention arm)
Procedure: Conventional (i.e. GTR) resection — Planned resection of ≥95% of the GAD-enhancing regions of tumor without expanding the resection beyond this margin.
  Arms: Conventional (i.e. GTR) resection

SUMMARY:
G-SUMIT is a pilot, phase II,randomized controlled trial to evaluate the feasibility of performing a large-scale trial in patients undergoing surgery for first-time diagnosis of high grade glioma (HGG) in a surgically favorable anatomical location to answer the following:

Does extending the margin of resection 1 cm beyond visible enhanced volume on MRI result in (a) an increase in overall survival? (b) result in a similar rate of "clinically-significant" neurological worsening during 30 days post surgery and quality of life at 6 and 12 months?

DETAILED DESCRIPTION:
This pilot, multi-centre, pragmatic randomized controlled trial is planned to simulate all aspects of a larger definitive trial comparing conventional versus supramarginal tumor resection at the time of the first surgical resection of HGG in appropriately selected patients. This pilot will help determine the ability to meet pre-specified criteria in identification, recruitment, and patient allocation, allow for refinement of eligibility criteria for optimal recruitment, confirm safety of procedure and ability to retain participants for the duration of the trial. Preliminary efficacy data will inform sample size calculations and estimation of resources required for the envisioned larger definitive trial.

ELIGIBILITY:
Inclusion Criteria:

1. Radiographic evidence of a GAD-enhancing intra-axial tumor consistent with HGG;
2. Age ≥18 ≤ 85 years;
3. Karnofsky Performance Score ≥ 60;
4. Location of tumor in a safe anatomical location and
5. Patient or substitute decision maker (SDM) able to understand and consent to study participation.

Exclusion Criteria:

1. Multi-focal tumor, gliomatosis cerebri (≥3 lobes of the brain affected), tumors crossing the midline, or leptomeningeal enhancement;
2. Previous craniotomy for tumor excision (stereotactic biopsy is permitted);
3. Known metastatic cancer;
4. Uncorrectable coagulopathy;
5. Unable to obtain GAD-enhanced brain MRI.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Enrollment | Collected at time of randomization, through end of enrollment period (2 years)
  The number of patients enrolled and successfully allocated to the intervention versus the control treatment

SECONDARY OUTCOMES:
Feasibility using eligibility | Screening/Enrollment
  Measures feasibility. Among all screened patients, the proportion of patients who meet the eligibility criteria
Feasibility using proportion of consent | Screening/Enrollment
  Measures feasibility. Among all screened patients, the proportion of patients consenting to participate
Feasibility using number of completed visits | Through study completion, on average 2 years
  Measures feasibility. Among all screened patients, the proportion of patients completing all scheduled follow-up assessments
Feasibility using Gross Total Resection | 2 days (+/- 1 day) post surgery
  Measures feasibility. The proportion of radiographically-confirmed gross total resection of contrast-enhancing tumor based on the first MRI after surgery.
Efficacy using overall survival | 6 weeks (+/- 2 weeks), 6 months (+/- 2 weeks) and 12 (+/- 1) months post surgery
  Measures efficacy. The date of death will be obtained from hospital records, outpatient follow up clinic notes, or provincial cancer registries.
Efficacy using progression-free survival | 6 weeks (+/- 2 weeks), 6 months (+/- 2 weeks) and 12 (+/- 1) months post surgery
  Measures efficacy. Assessment of progression-free survival based on the Modified Criteria for Radiographic Response Assessment in Glioblastoma (mRANO) criteria. The date of death will be obtained from hospital records, outpatient follow up clinic notes, or provincial cancer registries. Progression-free survival will be measured based on mRANO criteria during regular 3-month interval clinical and MRI follow up
Safety using neurological function | 2 (+/- 1) days and 6 weeks (+/- 2 weeks), days post surgery
  The NIH Stroke Scale (NIHSS) will be used to assess neurological function. The NIHSS is a validated neurologically-specific outcome tool originally developed for rapid grading of stroke symptoms adopted in surgical clinical trials as well.
Safety using global disability | 6 months (+/- 2 weeks) and 12 (+/- 1) months post surgery
  The modified rankin scale (mRS ) is a measure of global disability that has been widely used to assess outcome after stroke.
  The scale consists of six grades from 0 (no symptoms) to 5 (severe disability); 6 indicates death.
Safety using quality of life | 6 months (+/- 2 weeks) and 12 (+/- 4 weeks) post surgery, 24 (+/- 4 weeks) post surgery
  The overall quality of life will be assessed either in-person or over the phone using the EuroQol-5 (EQ-5D). The EQ-5D is a generic instrument used to measure quality of life, designed for self-completion by respondents either face-to-face or over telephone interview, also available in proxy version through care giver.
Safety using 6 weeks (+/- 2 weeks) all cause-mortality | 6 weeks (+/- 2 weeks) post surgery
  Will collect mortality data.
Radiological | 2 (+/- 1) days, 6 months (+/- 2 weeks) and 12 (+/- 1) months
  Volumetric measurement of contrast enhancement on MRI

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Pirouzmand, MD, MSc, FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre; Alireza Mansouri, MD MSc FRCSC, Principal Investigator — Penn State Cancer Institute; Damon Scales, MD, PhD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (6):
- The Pennsylvania State University, University Park, Pennsylvania, United States
- Canada (5):
  - Mackenzie Health Sciences Center, Edmonton, Alberta
  - Kingston Health Sciences Centre, Kingston, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Mansouri A, Lai C, Scales D, Pirouzmand F. A phase II pilot randomized controlled trial to assess the feasibility of the "supra-marginal" surgical resection of malignant glioma (G-SUMIT: Glioma supra marginal incision trial) study protocol. Pilot Feasibility Stud. 2022 Jul 5;8(1):138. doi: 10.1186/s40814-022-01104-1. PMID 35791008